CLINICAL TRIAL: NCT06489990
Title: Implementation Research on the Intervention Mode of " Comorbidity-Co-causes-Joint-prevention" Comprehensive Demonstration District of Depression and Obesity Among Children and Adolescents in Beijing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Peking University (Other); Center for Disease Control and Prevention of Bejing Economic-Technoloogical Develeopment Area (Unknown)
Responsible Party: Principal Investigator, Linghui Meng, Director of Department of Clinical Research Methodology，Beijing Anding Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CFH2024-1G-2121
Record Dates: First submitted 2024-06-12; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Depression; Obesity; High Risk of Depression; Overweight
Keywords: children; adolescents; depression; obesity; effectiveness evaluation; intervention mode
MeSH Terms: conditions — Depression; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): the intervention is combination intervention strategy of " Comorbidity-Co-causes-Joint-prevention"
  Interventions: Combination Product: combination intervention strategy of [Comorbidity-Co-causes-Joint-prevention]
- control group (Placebo Comparator): receiving routine health education and mental health knowledge
  Interventions: Combination Product: routine health education and mental health knowledge

INTERVENTIONS:
Combination Product: combination intervention strategy of [Comorbidity-Co-causes-Joint-prevention] — combination intervention strategy of [Comorbidity-Co-causes-Joint-prevention]
  Arms: intervention group
Combination Product: routine health education and mental health knowledge — routine health education and mental health knowledge
  Arms: control group

SUMMARY:
Depression and obesity have become the most prominent health problems among adolescents and have caused a heavy burden on the health and social economy of the whole population. There are high incidence, comorbidity and co-pathogenic factors of depression and obesity in adolescents, but there is still a lack of research on joint prevention strategies and multi-sectoral collaborative prevention and control network. This project plans to screen and integrate effective intervention measures based on multi-stage optimization strategy, developing an intervention mode of [Comorbidity-Co-causes-Joint-prevention] for adolescents with depression or/and obesity, and then carry out with children or adolescents in Beijing based on digital platform. The investigators will be considering the accessibility, sustainability and replicability of the implement based on the RE-AIM framework including the coverage of population and organizations as well as the effect, implement and sustainability of the interventions. The research will be promoted with the help of the National Clinical Research Center for Mental Disorders and Monitoring of Student Common Diseases and Health Influencing Factors. The results of the research will establish an intervention mode of [Comorbidity-Co-causes-Joint-prevention] and a promotion model for adolescents' depression and obesity in Beijing, providing support for the realization of Healthy China 2030 and Healthy Beijing 2030 Plans.

ELIGIBILITY:
Inclusion Criteria:

* Stage I (screening stage):

  1. Middle school students in Beijing Economic-Technological Development Area and other districts of Beijing, both male and female;
  2. Students themselves and their guardians are willing to participate in this study and sign written informed consent file.

     Stage Ⅱ:

     Middle school students who were identified as high risk of depression and/or obesity in Stage I in Beijing Economic-Technological Development Area and other districts of Beijing, the screening criteria are as follows:

     ① CES-DC score ≥16 points;

     ② BMI ≥WS/T586-2018: Screened as overweight and obesity among school-age children and adolescents, according to the recommendation by the National Health Commission;

     ③ Students themselves and their guardians are willing to participate in this study and provide written informed consent.

     Exclusion Criteria:
* Stage I:

  1. Having serious physical or genetic disease that is not suitable for participation in the study;
  2. Have been evaluated that not suitable for this study by investigators.

Stage Ⅱ:

1. Having serious physical or genetic disease that is not suitable for participation in the study;
2. Have been evaluated that not suitable for this study by investigators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9(PHQ-9) | From enrollment to the end of treatment at baseline、12weeks、6months
  The score ranges from 0 to 27, the higher scores mean more serious depression

SECONDARY OUTCOMES:
BMI | From enrollment to the end of treatment at baseline、12 weeks、6months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anding Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Gui P, Lin J, Zhao Y, Zhang X, Song Y, Meng L. Implementation research on the intervention mode of "Comorbidity-Co-causes-Joint-prevention" comprehensive demonstration district of depression and obesity among children and adolescents in Beijing: study protocol. BMC Public Health. 2025 Sep 30;25(1):3232. doi: 10.1186/s12889-025-24339-y. PMID 41029633